CLINICAL TRIAL: NCT02839499
Title: Screening of Obstructive Sleep Apnea Syndrome in Residents of a Unit of Long-term Care Under Mixed Food
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: physician's departure
Sponsor: Centre Hospitalier Universitaire de Saint Etienne (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 1608080; 2016-A01066-45 (Other: ANSM)
Record Dates: First submitted 2016-07-08; First posted 2016-07-21 (Estimated); Last update posted 2019-03-21 (Actual); Status verified 2019-03

CONDITIONS: Obstructive Sleep Apnea Syndrome
Keywords: seniors; mixed food; normal texture food
MeSH Terms: conditions — Sleep Apnea, Obstructive | interventions — Activities of Daily Living

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- mixed food (Experimental): experimental group with RU sleeping®, autonomy scale (ADL and AGGIR) and various activity scale (IADL)
  Interventions: Device: RU sleeping®; Other: autonomy scale (ADL and AGGIR); Other: various activity scale (IADL)
- normal texture food (Other): control group with RU sleeping®, autonomy scale (ADL and AGGIR) and various activity scale (IADL)
  Interventions: Device: RU sleeping®; Other: autonomy scale (ADL and AGGIR); Other: various activity scale (IADL)

INTERVENTIONS:
Device: RU sleeping® — Each patient included in the study has a test by RU-sleeping. The diagnosis of obstructive sleep apnea syndrome will be asked for an index of respiratory events estimated as greater than or equal to 10.
Other: autonomy scale (ADL and AGGIR) — autonomy data
Other: various activity scale (IADL) — activity of life data

SUMMARY:
Obstructive sleep apnea is a condition that affects 40% to 62% of the population aged over 60 years with major consequences especially on the cardiovascular system.

This syndrome consists of a staff of the pharyngeal muscles. These muscles are also involved in swallowing phenomena and chews, or many elderly patients are subjected to a mixed diet, logically leading to atrophy of the muscles aerodigestive crossroads.

Muscle wasting ENT induced a mixed food could promote collapsibility of VAS, exposing the individual to a higher risk of apnea and hypopnea during sleep.

The objective of this study is to determine if there is a significant increase in the prevalence of obstructive sleep apnea syndrome in the elderly patients residing in long term care units, receiving a mixed food compared to residents in supply to normal texture.

ELIGIBILITY:
Inclusion Criteria:

* Resident of a unit of long-term care
* Recipient or affiliated with Social Security
* Signature of consent by the patient, guardian or person of trust

and mixed food or normal texture food

Exclusion Criteria:

* OSA diagnosed and treated earlier
* Patients with an abnormal upper airway out edentation
* Patients unable to give informed consent and having no confidence in individual capacity to do so.
* Patients with a gastrostomy or jejunostomy

Min Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 39 (Actual)
Dates: Start 2016-11-15 (Actual); Primary Completion 2017-03-01 (Actual); Study Completion 2017-03-01 (Actual)

PRIMARY OUTCOMES:
measure of the index of respiratory events | up to 24 hours
  measured with holter (RU-sleeping®)

CONTACTS AND LOCATIONS:
Overall Officials: Emilie CRAWFORD-ACHOUR, MD, Principal Investigator — CHU de Saint Etienne
Locations (1):
- CHU de Saint Etienne, Saint-Etienne, France

IPD SHARING:
Plan to Share IPD: No